CLINICAL TRIAL: NCT03397745
Title: Which Bispectral Index Score is Reliable Throughout Esophageal Cancer Operation?
Brief Title: Bispectral Index Throughout Esophageal Cancer Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMC2017-12-033
Record Dates: First submitted 2018-01-02; First posted 2018-01-12 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer
Keywords: bispectral index; lateral decubitus position; one lung ventilation
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIS group (Other): Patients who received the esophageal surgery
  Interventions: Device: BIS

INTERVENTIONS:
Device: BIS — All patients applied BIS on both side (Left and Right)

SUMMARY:
The investigators try to conduct a study to assess the impact of changing patients' lateral decubitus position on BIS readings during esophageal cancer operation. Also, the investigators evaluate the effects of one-lung ventilation and total lung ventilation on BIS value with inhalation agent.

DETAILED DESCRIPTION:
Bispectral index (BIS) was developed to monitor a patient's level of consciousness under general anesthesia. Several factors have been found to alter BIS readings without affecting the depth of anesthesia.Changing a patient's position (head up and head down) significantly affects the BIS values, which might affect the interpretation of anesthetic depth.

During esophageal cancer surgery, there were several factors which could affect to BIS values.First, the surgical positions are consisted with supine and lateral decubitus position more than 1 h. Thus, the investigators compare the BIS value of both side on supine and lateral decubitus position by both side approach. Second, the one lung ventilation was applied for surgical filed. It alters the oxygenation and the cerebral flow. Because of these effects, the BIS monitoring can differ by the period of surgery. Thus, in this study, the BIS value of both side monitor throughout the surgery.

ELIGIBILITY:
Inclusion Criteria:

the patients who are planned the esophageal cancer operation

Exclusion Criteria:

* patient who has dermatitis
* patient who refuse to participate in this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Change in Bispectral index score | after lateral decubitus position 5 mins, 10 mins, 20 mins, 30 mins
  The difference of both side BIS value on lateral decubitus position

SECONDARY OUTCOMES:
the asymmetry of BIS | after supine position 5 mins, 10 mins, 20 mins, 30 mins
  The difference of BIS on supine position
oxygenation and BIS | intraoperative
  the effects of arterial blood gas analysis (O2 mmH2O and CO2 mmH2O) on BIS
The changes of BIS | intraoperative
  the difference of BIS divided to 3 BIS level ( <40,40-60,>60)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No